CLINICAL TRIAL: NCT05488067
Title: The Safety and Efficacy of Atorvastatin on Xanthoma in Alagille Syndrome
Brief Title: Atorvastatin Therapy on Xanthoma in Alagille Syndrome
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATO-ALGS-XAN
Record Dates: First submitted 2022-08-01; First posted 2022-08-04 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Alagille Syndrome; Atorvastatin; Xanthoma
MeSH Terms: conditions — Alagille Syndrome; Xanthomatosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Atorvastatin+ALGS-Xanthoma (Experimental): Drug: atorvastatin Dosage form: tablet Route of administration: oral Duration: 6 months （After 6 months of medication, according to the actual situation of the patient, choose to maintain the original dosage, gradually reduce the dosage or stop the medication）
  Administration method:
  Initial dose: ① < 1 year old: 1.25mg/d, qd; ② 1-5 years old: 2.5mg/d, qd; ③ 6-9 years old: 5mg/d, qd; ④ ≥ 10 years old: 10mg/d, qd. The maximum dose is 40mg/d and not more than 1mg/kg/d. During the follow-up, the medication was adjusted according to the laboratory results until non-HDL-C≤4.2mmol/L（162 mg/dL）, xanthoma disappear, or the patient had moderate or more serious adverse reactions.
  Interventions: Drug: atorvastatin

INTERVENTIONS:
Drug: atorvastatin — Oral atorvastatin treatment for ALGS children with xanthoma
  Other Names: Lipitor

SUMMARY:
To observe the efficacy and safety of atorvastatin on xanthoma in Alagille syndrome through a prospective study.

DETAILED DESCRIPTION:
Alagille syndrome (ALGS, OMIM 118450) is an important cause of chronic cholestasis in children, and the incidence rate is about 1:30000~1:50000. Most patients with ALGS have hypercholesterolemia. In severe cases, multiple xanthomas can be seen, and some patients are accompanied by severe itching and pain. Disfigured xanthomas affect the normal social interaction of patients, thereby causing physical and mental damage to children. At present, xanthoma caused by hypercholesterolemia can be cured by treating the primary disease, taking lipid-lowering drugs (such as bile acid chelators, ezetimibe, statins, etc.), or lipoprotein apheresis. If it affects the beauty or function, local treatment such as 33% trichloroacetic acid dot coating, carbon dioxide laser, liquid nitrogen freezing or surgical resection is feasible, and even surgical operation( such as portal vena cava anastomosis, liver transplantation). Compared with expensive lipoprotein apheresis and other invasive therapies, taking lipid-lowering drug has the advantages of higher acceptance, lower cost and higher safety. However, at present, there are no guidelines for application of oral lipid-lowering drugs in children under 6 years old with hypercholesterolemia. Therefore, the purpose of this study is to clarify the safety and efficacy of atorvastatin on xanthoma in ALGS , so as to provide reference for the treatment of ALGS patients' xanthomas.

Risk prevention and treatment: The patients began to take atorvastatin from a small dose, followed up closely in the early stage (2-4 weeks) to see if the patients had obvious discomfort such as myalgia, and monitored the changes of Biochemistry (CK, ALT, AST, etc.). If moderate or more serious adverse reactions occurred during the trial or the following laboratory abnormalities occurred (CK exceeded 10 times the upper limit of normal; ALT or AST had been continued to rise, exceeding 2 times the baseline value), atorvastatin was temporarily stopped, and patients should be rechecked within 2 weeks. It is necessary to reevaluate and decide whether to restart atorvastatin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet the ALGS diagnostic criteria;
* Xanthoma of skin;
* Before treatment with atorvastatin,non-HDL-C≥5.76mmol/L（223 mg/dL）;
* Informed consent;
* Age 0-17 years old, male or female;
* Taking bile acid chelator (colenemide) has no obvious effect or intolerance.

Exclusion Criteria:

* Liver transplantation has been performed;
* In the recovery period of cholestasis, xanthoma is obviously subsiding;
* Patients with serious systemic diseases and unstable vital signs;
* Progressive active liver injury, such as continuous increase of transaminase;
* Serious myopathy;
* Known to be allergic to any component of atorvastatin;
* The weight is less than 5kg.

Ages: 1 Day to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-03-22 (Estimated); Study Completion 2025-03-22 (Estimated)

PRIMARY OUTCOMES:
Grade change of xanthoma | from enrollment to the 3th/6th month
  The grade change of xanthoma would be assessed at the 3th/6th month after enrollment 【Explanation：Xanthomas were graded as 0 = none, 1 = minimal, 2 =moderate, 3 = disfiguring, and 4 = disabling. Minimal xanthomas signified fewer than 20 scattered individual lesions, moderate represented more than 20 lesions that did not interfere with or limit activities, disfiguring represented large numbers of lesions that by their large numbers or size caused distortion of the face or xtremities, and disabling signified that the xanthomas interfered with function (such as hand use or ability to walk) because of excess size or number.】

SECONDARY OUTCOMES:
non-HDL-C change | from enrollment to the 3th/6th month
  The non-HDL-C change would be measured at the 3th/6th month after enrollment 【Explanation: non-HDL-C is defined as the difference between total cholesterol and HDL-C】
Incidence of adverse events | from enrollment to the 3th/6th month
  It is a binary variable. Incidence Rates for adverse event（including：rhabdomyolysis and myopathy，liver enzymes exceeded twice the baseline value，nasopharyngitis, muscle pain，diarrhea，nausea, fever，urinary tract infection, joint swelling，epistaxis，urticaria，etc.）would be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gilbert MA, Bauer RC, Rajagopalan R, Grochowski CM, Chao G, McEldrew D, Nassur JA, Rand EB, Krock BL, Kamath BM, Krantz ID, Piccoli DA, Loomes KM, Spinner NB. Alagille syndrome mutation update: Comprehensive overview of JAG1 and NOTCH2 mutation frequencies and insight into missense variant classification. Hum Mutat. 2019 Dec;40(12):2197-2220. doi: 10.1002/humu.23879. Epub 2019 Aug 26. PMID 31343788
- [Background] Ben Ameur S, Chabchoub I, Telmoudi J, Belfitouri Y, Rebah O, Lacaille F, Aloulou H, Mehrzi A, Hachicha M. Management of cholestatic pruritus in children with Alagille syndrome: Case report and literature review. Arch Pediatr. 2016 Dec;23(12):1247-1250. doi: 10.1016/j.arcped.2016.09.004. Epub 2016 Oct 27. PMID 28492167
- [Background] Martinsen MH, Klausen IC, Tybjaerg-Hansen A, Hedegaard BS. Autosomal recessive hypercholesterolemia in a kindred of Syrian ancestry. J Clin Lipidol. 2020 Jul-Aug;14(4):419-424. doi: 10.1016/j.jacl.2020.06.002. Epub 2020 Jun 8. PMID 32636080
- [Background] Lin M, Dai H, Zhao S. Long-term atorvastatin-ezetimibe-probucol triple therapy for homozygous familial hypercholesterolaemia from early childhood. Cardiol Young. 2016 Jan;26(1):197-201. doi: 10.1017/S1047951115000591. Epub 2015 Apr 24. PMID 25907359
- [Background] Sreedharan AV, Pek SLT, Tan TH, Tavintharan S, Yap F. Successful pharmacological management of a child with compound heterozygous familial hypercholesterolemia and review of the recent literature. J Clin Lipidol. 2020 Sep-Oct;14(5):639-645. doi: 10.1016/j.jacl.2020.07.006. Epub 2020 Jul 15. PMID 32800790
- [Background] Luirink IK, Hutten BA, Greber-Platzer S, Kolovou GD, Dann EJ, de Ferranti SD, Taylan C, Bruckert E, Saheb S, Oh J, Driemeyer J, Farnier M, Pape L, Schmitt CP, Novoa FJ, Maeser M, Masana L, Shahrani A, Wiegman A, Groothoff JW. Practice of lipoprotein apheresis and short-term efficacy in children with homozygous familial hypercholesterolemia: Data from an international registry. Atherosclerosis. 2020 Apr;299:24-31. doi: 10.1016/j.atherosclerosis.2020.01.031. Epub 2020 Feb 18. PMID 32199148
- [Background] Shurberg JL, Resnick RH, Koff RS, Ros E, Baum RA, Pallotta JA. Serum lipids, insulin, and glucagon after portacaval shunt in cirrhosis. Gastroenterology. 1977 Feb;72(2):301-4. PMID 830579
- [Background] Kakaei F, Nikeghbalian S, Kazemi K, Salahi H, Bahador A, Dehghani SM, Dehghani M, Nejatollahi SM, Shamsaeefar A, Khosravi MB, Malek-Hosseini SA. Liver transplantation for homozygous familial hypercholesterolemia: two case reports. Transplant Proc. 2009 Sep;41(7):2939-41. doi: 10.1016/j.transproceed.2009.07.028. PMID 19765481
- [Background] Larrosa-Haro A, Saenz-Rivera C, Gonzalez-Ortiz M, Coello-Ramirez P, Vazquez-Camacho G. Lack of cholesterol-lowering effect of graded doses of cholestyramine in children with Alagille syndrome: a pilot study. J Pediatr Gastroenterol Nutr. 2003 Jan;36(1):50-3. doi: 10.1097/00005176-200301000-00011. PMID 12499996
- [Background] Sheflin-Findling S, Arnon R, Lee S, Chu J, Henderling F, Kerkar N, Iyer K. Partial internal biliary diversion for Alagille syndrome: case report and review of the literature. J Pediatr Surg. 2012 Jul;47(7):1453-6. doi: 10.1016/j.jpedsurg.2012.04.008. PMID 22813814
- [Background] Quek SC, Aw M, Quak SH, Prabhakaran K, Tan KC. Liver transplantation in a child with severe hypercholesterolaemia in Alagille syndrome. Ann Acad Med Singap. 2001 Jan;30(1):44-7. PMID 11242624
- [Background] Nakajima H, Tsuma Y, Fukuhara S, Kodo K. A Case of Infantile Alagille Syndrome With Severe Dyslipidemia: New Insight into Lipid Metabolism and Therapeutics. J Endocr Soc. 2022 Jan 18;6(3):bvac005. doi: 10.1210/jendso/bvac005. eCollection 2022 Mar 1. PMID 35155971
- [Background] Tapia Ceballos L, Picazo Angelin B, Ruiz Garcia C. [Use of statins in children]. An Pediatr (Barc). 2008 Apr;68(4):385-92. doi: 10.1157/13117712. Spanish. PMID 18394386
- [Background] Melvin AJ, Montepiedra G, Aaron L, Meyer WA 3rd, Spiegel HM, Borkowsky W, Abzug MJ, Best BM, Crain MJ, Borum PR, Graham B, Anthony P, Shin K, Siberry GK; P1063 Study Team. Safety and Efficacy of Atorvastatin in Human Immunodeficiency Virus-infected Children, Adolescents and Young Adults With Hyperlipidemia. Pediatr Infect Dis J. 2017 Jan;36(1):53-60. doi: 10.1097/INF.0000000000001352. PMID 27749649
- [Background] Hari P, Khandelwal P, Satpathy A, Hari S, Thergaonkar R, Lakshmy R, Sinha A, Bagga A. Effect of atorvastatin on dyslipidemia and carotid intima-media thickness in children with refractory nephrotic syndrome: a randomized controlled trial. Pediatr Nephrol. 2018 Dec;33(12):2299-2309. doi: 10.1007/s00467-018-4036-x. Epub 2018 Aug 8. PMID 30091061
- [Background] Langslet G, Breazna A, Drogari E. A 3-year study of atorvastatin in children and adolescents with heterozygous familial hypercholesterolemia. J Clin Lipidol. 2016 Sep-Oct;10(5):1153-1162.e3. doi: 10.1016/j.jacl.2016.05.010. Epub 2016 Jun 7. PMID 27678432
- [Background] Gandelman K, Glue P, Laskey R, Jones J, LaBadie R, Ose L. An eight-week trial investigating the efficacy and tolerability of atorvastatin for children and adolescents with heterozygous familial hypercholesterolemia. Pediatr Cardiol. 2011 Apr;32(4):433-41. doi: 10.1007/s00246-011-9885-z. Epub 2011 Jan 23. PMID 21259004
- [Background] Araujo MB, Pacce MS. A 10-year experience using combined lipid-lowering pharmacotherapy in children and adolescents. J Pediatr Endocrinol Metab. 2016 Nov 1;29(11):1285-1291. doi: 10.1515/jpem-2016-0117. PMID 27718491
- [Background] Niedra E, Chahal N, Manlhiot C, Yeung RS, McCrindle BW. Atorvastatin safety in Kawasaki disease patients with coronary artery aneurysms. Pediatr Cardiol. 2014 Jan;35(1):89-92. doi: 10.1007/s00246-013-0746-9. Epub 2013 Jul 18. PMID 23864222
- [Background] Tremoulet AH, Jain S, Jone PN, Best BM, Duxbury EH, Franco A, Printz B, Dominguez SR, Heizer H, Anderson MS, Glode MP, He F, Padilla RL, Shimizu C, Bainto E, Pancheri J, Cohen HJ, Whitin JC, Burns JC. Phase I/IIa Trial of Atorvastatin in Patients with Acute Kawasaki Disease with Coronary Artery Aneurysm. J Pediatr. 2019 Dec;215:107-117.e12. doi: 10.1016/j.jpeds.2019.07.064. Epub 2019 Sep 24. PMID 31561960
- [Background] Huang J, Li L, Zhang J, Gao C, Quan W, Tian Y, Sun J, Tian Q, Wang D, Dong J, Zhang J, Jiang R. Treatment of Relapsed Chronic Subdural Hematoma in Four Young Children with Atorvastatin and Low-dose Dexamethasone. Pharmacotherapy. 2019 Jul;39(7):783-789. doi: 10.1002/phar.2276. Epub 2019 May 28. PMID 31069819
- [Background] Agrawal D, Manchanda SC, Sawhney JPS, Kandpal B, Jain R, Mehta A, Mohanty A, Passey R, Makhija A, Sharma MK. To study the effect of high dose Atorvastatin 40mg versus 80mg in patients with dyslipidemia. Indian Heart J. 2018 Dec;70 Suppl 3(Suppl 3):S8-S12. doi: 10.1016/j.ihj.2018.01.034. Epub 2018 Jan 31. PMID 30595326